CLINICAL TRIAL: NCT00000383
Title: Treatment of PTSD in Sexually Abused Children
Brief Title: Treatment of Post-Traumatic Stress Disorder (PTSD) in Sexually Abused Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of Medicine and Dentistry of New Jersey (Other)
Responsible Party: Principal Investigator, Judith Cohen, Principal Investigator, Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R10MH055963 (NIH); 1R10MH055963 (NIH); 1R10MH056224 (NIH)
Record Dates: First submitted 1999-11-02; First posted 1999-11-03 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: Adolescence; Child; Cognitive Therapy; Comparative Study; Female; Human; Male; Stress Disorders, Post-Traumatic; Child Abuse, Sexual; Stress Disorders, Post-Traumatic -- *therapy; Child Abuse, Sexual -- *psychology
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Coitus; Stress Disorders, Traumatic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Trauma-Focused CBT (Experimental): Trauma -Focused CBT provides 12 sessions (45 minutes child, 45 minutes parent) of CBT treatment. This includes therapist-directed trauma-focused skills training, exposure, parenting, conjoint parent-child sessions, and safety component provided to child and parent.
  Interventions: Behavioral: Trauma-Focused CBT
- Child Centered Therapy (Active Comparator): Child Centered Therapy provides 12 sessions (45 minutes child, 45 minutes parent) of supportive interventions. This includes client-directed activities focused on the needs and interests of the child or parent, respectively.
  Interventions: Behavioral: Child-Centered Therapy

INTERVENTIONS:
Behavioral: Trauma-Focused CBT — Structured skills, exposure, trauma-specific interventions
  Other Names: TF-CBT
  Arms: Trauma-Focused CBT
Behavioral: Child-Centered Therapy — Client-directed supportive interventions
  Other Names: CCT
  Arms: Child Centered Therapy

SUMMARY:
The purpose of this study is to compare the effectiveness of two psychological therapies used to treat PTSD in children who have recently been sexually abused: Trauma-Focused Cognitive Behavioral Therapy (TF-CBT) vs Child Centered Therapy (CCT).

Child sexual abuse is a common experience that has serious mental health consequences, including the development of PTSD and other abuse-related problems.

All children will be assigned randomly (like tossing a coin) to receive either SAS-CBT or NST at each of two sites. In addition, the parents and the child will receive individual therapy for 12 weeks. The child will be monitored to evaluate his/her response to therapy. Assessments will take place before and just following treatment, and then 6 and 12 months post-treatment.

A child may be eligible for this study if he/she:

Has been sexually abused, is suffering from PTSD as a result of the abuse, and is 8 to 14 years old.

DETAILED DESCRIPTION:
To evaluate the comparative efficacy of Trauma-Focused Cognitive Behavioral Therapy (TF-CBT) vs Child Centered Therapy (CCT) in decreasing symptoms of Post-Traumatic Stress Disorder (PTSD) following recent sexual abuse.

Child sexual abuse is a common experience that has serious mental health consequences, including the development of PTSD and other abuse-related and general psychopathological symptoms.

Patients are randomly assigned to receive either TF-CBT or CCT at each of two sites, and will be provided with 12 weeks of individual therapy for children and parents. Treatment is monitored for compliance with the respective treatment models through intensive supervision, audiotaping of sessions, rating of sessions with use of adherence checklists, and independent blind rating of audiotapes. Treatment outcome is evaluated through the use of several self-, parent-, and teacher-report standardized instruments, administered at pre- and post-treatment, and follow-up evaluations at 6 and 12 months. The project also assesses differential treatment impact by gender and ethnicity, and attempts to evaluate the impact of specific components of the treatment process in mediating treatment outcome. Specifically, the project evaluates the differential effectiveness of the two treatment modalities in improving the subject's abuse-related attributions and perceptions, parenting practices, familial adaptability and cohesiveness, parent support, and parental emotional reaction to the abuse, and the impact of improving these variables on treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

-

Patients must have:

1. Post-Traumatic Stress Disorder (PTSD) symptoms (at least 5 with at least one symptom in each of 3 PTSD clusters) related to sexual abuse
2. Confirmed child sexual abuse history
3. Speak English
4. Parent willing to participate in treatment

Exclusion Criteria:

1. Active psychotic disorder resulting in inability to participate in CBT
2. Active substance abuse disorder that resulted in significant impairment 3 Serious developmental disorder precluding participation in CBT

4) If on psychotropic medication, not on stable dose for at least 4 weeks 5) Receiving ongoing psychotherapy outside of study

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 229 (Actual)
Dates: Start 1997-09; Primary Completion 2001-09 (Actual); Study Completion 2002-09 (Actual)

PRIMARY OUTCOMES:
PTSD | 12 weeks; 6- and 12- month follow-up
  Change in child PTSD total PTSD symptoms, PTSD cluster symptoms, PTSD diagnosis as measured by the K-SADS-PL

SECONDARY OUTCOMES:
Depression | 12 weeks; 6- and 12-month follow up
  Change in child depressive symptoms measured by the Child Depression Inventory
Anxiety | 12 weeks; 6 and 12-month follow-up
  Change in child anxiety symptoms measured by State Trait Anxiety Inventory
Maldaptive Cognitions | 12 weeks; 6 and 12 month follow-up
  Change in maladaptive trauma-related cognitions measured by the Children'sAttributions and Perceptions Scale
Shame | 12 weeks; 6 and 12 month follow up
  Change in child shame measured by SHAME scale
Parent depression | 12 weeks; 6 and 12 month follow up
  Change in parental depression measured by Beck Depression Inventory
Parent Emotional Distress | 12 weeks; 6 and 12 month follow up
  Change in parental distress related to child's abuse measured by Parental Emotional Reaction Questionnaire
Parental Support | 12 weeks; 6 and 12 month follow up
  Change in parental support of child measured by Parental Support Questionnaire
Positive Parenting Practices | 12 weeks; 6 and 12 month follow up
  Change in positive parenting measured by Parenting Practices Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Judith A. Cohen, MD, Principal Investigator — Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute); Esther Deblinger, PhD, Principal Investigator — University of Medicine and Dentistry of New Jersey
Locations (3):
- United States (3):
  - Center for Children's Support, University of Medicine and Dentistry - New Jersey, Stratford, New Jersey
  - Allegheny General Hospital Center for Traumatic Stress in Children and Adolescents, Pittsburgh, Pennsylvania
  - Center for Traumatic Stress in Children & Adolescents, Allegheny General Hospital, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Cohen JA, Deblinger E, Mannarino AP, Steer RA. A multisite, randomized controlled trial for children with sexual abuse-related PTSD symptoms. J Am Acad Child Adolesc Psychiatry. 2004 Apr;43(4):393-402. doi: 10.1097/00004583-200404000-00005. PMID 15187799